CLINICAL TRIAL: NCT02573493
Title: Phase II Non-Randomized Three Arm Trial of Induction Chemotherapy With Nab-Paclitaxel and Cisplatin (AP: Arms 1 and 3) or Single Agent Nab-paclitaxel (A: Arm 2) as Induction Therapy Followed by Definitive Concurrent Chemoradiation for Locally Advanced Squamous Cell Carcinoma of the Head and Neck (HNSCC): "The APA Trial".
Brief Title: Nab-Paclitaxel and Cisplatin or Nab-paclitaxel as Induction Therapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Acronym: APA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201510013
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Carcinoma, Squamous Cell of the Head and Neck; Cancer of Head and Neck; Cancer of the Head and Neck; Head and Neck Cancer; Neoplasms, Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Cisplatin; Cetuximab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: nab-Paclitaxel and cisplatin (AP) + CRT (Experimental): * Six weeks of nab-paclitaxel (100 mg/m2/week) and cisplatin (75 mg/m2 days 1 and 22) followed by primary tumor site (PTS) assessment
  * If complete response (CR)/partial response (PR), three more weeks of nab-paclitaxel and cisplatin followed by concurrent chemoradiation therapy (CRT)
  * If <PR, move directly to CRT if not surgical candidates.
  * CRT includes cisplatin which will begin 1 to 35 days after the completion of cycle 3. The first dose of cisplatin will be given during the initial 5 days of definitive radiation therapy, the second on approximately Day 22 of radiation, and the third on approximately Day 43 of radiation.
  * It is strongly recommended that intensity-modulated radiation therapy (IMRT) begin within 21 to 42 days (no later than 56 days) after the start of cycle 3. The total dose will be 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to areas considered to be an intermediate risk.
  Interventions: Drug: nab-Paclitaxel; Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy
- Arm 2: nab-Paclitaxel (A) + CRT (Experimental): * Six weeks of nab-paclitaxel (100 mg/m2/week) followed by primary tumor site (PTS) assessment
  * If CR/PR, three more weeks of nab-paclitaxel followed by CRT
  * If <PR, move directly to CRT if not surgical candidates.
  * CRT includes cetuximab and will begin 1 to 35 days after completion of cycle -Cetuximab will be started 7 days before starting definitive radiation therapy. The initial loading dose of cetuximab will be 400 mg/m^2. Subsequently, cetuximab will be given weekly at a dose of 250 mg/m^2 for seven additional doses concurrently with radiation therapy.
  * It is strongly recommended that IMRT begin within 21 to 42 days (no later than 56 days) after the start of cycle 3. The total dose will be 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to areas considered to be an intermediate risk.
  Interventions: Drug: nab-Paclitaxel; Biological: Cetuximab; Radiation: Intensity-Modulated Radiation Therapy
- Arm 3: nab-Paclitaxel and cisplatin (AP) + modified CRT (Experimental): * 6 weeks of nab-paclitaxel and cisplatin (days 1 & 22) followed by primary tumor site assessment
  * If CR/PR, cycle 3 of induction then 42Gy radiation, 1 dose of cisplatin or 6 doses cetuximab
  * If SD/PD: undergo surgery if candidate followed by CRT with 42 Gy RT and abbreviated cisplatin or cetuximab or 70Gy RT and 3 cycles of cisplatin or 8 doses of cetuximab
  * CRT includes Cisplatin and will begin 1-35 days after the completion of Cycle 3 of induction. Cisplatin will be given as 1 dose during the initial 5 days of definitive radiation therapy
  * Strongly recommended that radiation therapy begin within 28-49 days (and no later than 56 days) after the start of Cycle 3. Intensity modulated radiation therapy is to be used exclusively for this study.
  Interventions: Drug: nab-Paclitaxel; Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy

INTERVENTIONS:
Drug: nab-Paclitaxel
  Other Names: Abraxane
Drug: Cisplatin
  Other Names: cis-DDP; cis-Platinum II; cis-Diamminedichloroplatinum; DDP
  Arms: Arm 1: nab-Paclitaxel and cisplatin (AP) + CRT; Arm 3: nab-Paclitaxel and cisplatin (AP) + modified CRT
Biological: Cetuximab
  Other Names: Erbitux®
  Arms: Arm 2: nab-Paclitaxel (A) + CRT
Radiation: Intensity-Modulated Radiation Therapy
  Other Names: IMRT

SUMMARY:
In this trial, the objectives are to determine the efficacy and toxicity of induction chemotherapy (IC) with nab-paclitaxel + cisplatin (Arm 1: AP) and with nab-paclitaxel (Arm 2: A) alone in patients with HNSCC, and to compare these data to nab-paclitaxel, cisplatin, and 5-FU (APF). The investigators also hypothesize that the high anti-tumor efficacy of nab-paclitaxel in HNSCC is due to the upregulation of macropinocytosis, a result of the frequent presence of Ras and PI3K (and epidermal growth factor receptor -EGFR) activation in this cancer.

Amendment to Add Arm 3:

In this amendment, the investigators retain the AP + concurrent chemoradiation therapy (CRT) backbone but de-escalate the dose of radiation therapy (RT) from 70 Gy to 42 Gy. The investigators also plan to administer one dose (vs three) of cisplatin during RT. This novel treatment approach will be evaluated in patients with HPV-related oropharyngeal squamous cell carcinoma (OPSCC) (Arm 3), a sub-group with a very favorable prognosis.

ELIGIBILITY:
Inclusion Criteria: Arms 1 and 3 - AP

* Diagnosis of selected Stage III or IVa/b HNSCC. Arm 1: T2-T4 primary tumors. Arm 3: T2T1-T4 primary tumors. Although most of these patients will have regional nodal disease, patients with no nodal disease will also be eligible.
* Arm 1: Presence of disease at the oropharynx, hypopharynx, or larynx sub-sites.
* Arm 3: Presence of disease at the oropharynx sub-sites, which is HPV-related as verified by p16, a surrogate marker of HPV, or HPV ISH or PCR.
* Presence of measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan.
* At least 18 years of age.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 3 months after completing treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB-approved written informed consent document.
* ECOG performance status ≤ 1.
* Adequate bone marrow and organ function as defined below:

  * ANC: ≥ 1500/mcL.
  * Platelets: > 100,000/mcL.
  * Hemoglobin > 9.0 g/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * AST/ALT/alkaline phosphatase: ≤ 2.5 x ULN.
  * Serum creatinine: < 1.5 mg/dL or calculated GFR ≥ 75 cc/min. CrCl by Cockcroft Gault will be used to estimate GFR.
  * Pulmonary: no requirement for supplemental oxygen and no evidence of moderate-severe chronic obstructive pulmonary disease (COPD) by pulmonary function tests (PFTs).

Inclusion Criteria: Arm 2 - A

* Diagnosis of selected Stage III or IVa/b HNSCC. T2-T4 primary tumors. (Patients with T1 tumors will be excluded). Although most of these patients will have regional nodal disease, patients with no nodal disease will also be eligible.
* Presence of disease at the oropharynx, hypopharynx, or larynx sub-sites.
* Presence of measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan.
* At least 18 years of age.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 3 months after completing treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB-approved written informed consent document.
* ECOG performance status < 3.
* Adequate bone marrow and organ function as defined below:

  * ANC: ≥ 1500/mcL.
  * Platelets: ≥ 100,000/mcL.
  * Hemoglobin > 9.0 g/dL
  * Total bilirubin ≤ 2.0 mg/dL
  * AST/ALT/alkaline phosphatase: ≤ 5x ULN.
  * Calculated GFR >30 cc/min. CrCl by Cockcroft Gault will be used to estimate GFR.
  * Pulmonary: patients with a requirement for supplemental oxygen or evidence of moderate-severe COPD by PFTs are permitted to enroll.
* If a patient fully meets criteria for Arm 1, but has profound hearing loss and the physician feels that the patient should not receive Cisplatin, the patient will be eligible for Arm 2.
* If a patient fully meets criteria for Arm 1, but has a history of solid organ or bone marrow transplant, the patient will be eligible for Arm 2 (due to contraindications of Cisplatin with medications the patient is taking due to the transplant).

Exclusion Criteria (Arm 1 and Arm 2)

* Prior chemotherapy, prior EGFR targeted therapy, or prior radiation therapy for HNSCC.
* Disease at the nasopharyngeal, sinus, oral cavity, or other sub-site not specified as eligible.
* Diagnosis of unknown primary squamous cell carcinoma of the head and neck.
* History of prior invasive malignancy diagnosed within 3 years prior to study enrollment; exceptions are malignancies with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) that were treated with an expected curative outcome, such as squamous cell carcinoma of the skin, in-situ carcinoma of the cervix uteri, non-melanomatous skin cancer, carcinoma in situ of the breast, or incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
* Receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the agents used in this study.
* Taking cimetidine or allopurinol. If currently taking either of these medications, patient must discontinue for one week before receiving treatment with nab-paclitaxel.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or serious psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. A negative serum or urine pregnancy test is required at screening for all female patients of childbearing potential.
* Known to be HIV-positive on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with the study agents. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Peripheral neuropathy > grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Washington University School of Medicine, St Louis, Missouri
  - Sanford Cancer Center, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oppelt P, Ley J, Daly M, Rich J, Paniello R, Jackson RS, Pipkorn P, Liu J, Gay H, Palka K, Neupane P, Powell S, Spanos WC, Gitau M, Zevallos J, Thorstad W, Adkins D. nab-Paclitaxel and cisplatin followed by cisplatin and radiation (Arm 1) and nab-paclitaxel followed by cetuximab and radiation (Arm 2) for locally advanced head and neck squamous-cell carcinoma: a multicenter, non-randomized phase 2 trial. Med Oncol. 2021 Mar 8;38(4):35. doi: 10.1007/s12032-021-01479-w. PMID 33683482
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT: * Six weeks of nab-paclitaxel (100 mg/m2/week) and cisplatin (75 mg/m2 days 1 and 22) followed by primary tumor site (PTS) assessment
  * If complete response (CR)/partial response (PR), three more weeks of nab-paclitaxel and cisplatin followed by concurrent chemoradiation therapy (CRT)
  * If <PR, move directly to CRT if not surgical candidates.
  * CRT includes cisplatin (if cannot receive cisplain will receive cetuximab) which will begin 1 to 35 days after the completion of cycle 3. The first dose of cisplatin will be given during the initial 5 days of definitive radiation therapy, the second on approximately Day 22 of radiation, and the third on approximately Day 43 of radiation.
  * It is strongly recommended that intensity-modulated radiation therapy (IMRT) begin within 21 to 42 days (no later than 56 days) after the start of cycle 3. The total dose will be 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to areas considered to be an intermediate risk.
- Not Enrolled in Any Arm: -Determined to be not eligible after enrollment to study and was therefore not enrolled on any study arm.
Period: Overall Study
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT | Not Enrolled in Any Arm
Started | 40 | 40 | 15 | 1
Completed | 40 | 40 | 15 | 0
Not Completed | 0 | 0 | 0 | 1
Not completed — Determined to not be eligible after enrollment | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT: * Six weeks of nab-paclitaxel (100 mg/m2/week) and cisplatin (75 mg/m2 days 1 and 22) followed by primary tumor site (PTS) assessment
  * If complete response (CR)/partial response (PR), three more weeks of nab-paclitaxel and cisplatin followed by concurrent chemoradiation therapy (CRT)
  * If <PR, move directly to CRT if not surgical candidates.
  * CRT includes cisplatin (if cannot receive cisplatin will receive cetuximab) which will begin 1 to 35 days after the completion of cycle 3. The first dose of cisplatin will be given during the initial 5 days of definitive radiation therapy, the second on approximately Day 22 of radiation, and the third on approximately Day 43 of radiation.
  * It is strongly recommended that intensity-modulated radiation therapy (IMRT) begin within 21 to 42 days (no later than 56 days) after the start of cycle 3. The total dose will be 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to areas considered to be an intermediate risk.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT | Not Enrolled in Any Arm | Total
Number analyzed (Participants) | 40 | 40 | 15 | 1 | 96
Age, Continuous [Median (Full Range); unit: years] | 57.5 [42 to 77] | 65.5 [48 to 83] | 61 [41 to 68] | 62 [62 to 62] | 61 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 1 | 1 | 14
  Male | 36 | 32 | 14 | 0 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 39 | 15 | 1 | 95
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 3 | 0 | 0 | 11
  White | 32 | 37 | 15 | 1 | 85
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 15 | 1 | 96

OUTCOME MEASURES:

1. Primary Outcome: Arm 1 and Arm 2: Clinical Complete Response Rate as Measured by Clinical Exam at the Primary Tumor Site
Description: * Assessment of primary tumor site will be done by laryngoscopy performed in the office or in the operating room. The primary tumor response to the first two cycles of induction will be assessed using visual categorical response. The percent change from baseline will be dictated in the ear, nose, and throat (ENT) physician's clinical exam note.
  * Complete response = complete resolution - 100% decrease/minimal residual mucosal abnormality
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Population: Only participants enrolled in Arm 1 and Arm 2 are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 0
Participants | 28 | 8 |

2. Primary Outcome: Arm 3: Median Percent Weight Loss
Time Frame: Completion of treatment (estimated to be 11-15 weeks)
Population: Only participants enrolled in Arm 3 are evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of weight loss
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 0 | 0 | 15
percentage of weight loss |  |  | 6.7 [2.2 to 12.9]

3. Secondary Outcome: Arms 1, 2, and 3: Clinical Partial Response Rate as Measured by Clinical Exam at the Primary Tumor Site
Description: * Assessment of primary tumor site will be done by laryngoscopy performed in the office or in the operating room. The primary tumor response to the first two cycles of induction will be assessed using visual categorical response. The percent change from baseline will be dictated in the ENT physician's clinical exam note.
  * Partial response - 99-50% decrease
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 15
Participants | 11 | 28 | 6

4. Secondary Outcome: Arms 1, 2 and 3: Clinical Complete Response Rate as Measured by Clinical Exam at the Involved Regional Nodes
Description: * The involved neck node response to the first two cycles of induction will be assessed using visual categorical response. The neck node measurements will be performed clinically by the treating medical oncology physician and dictated in his/her assessment note.
  * Complete response - complete resolution - 100% decrease/minimal residual mucosal abnormality
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 30 | 33 | 11
Participants | 18 | 14 | 3

5. Secondary Outcome: Arms 1, 2, and 3: Clinical Partial Response Rate as Measured by Clinical Exam at the Involved Regional Nodes
Description: * The involved neck node response to the first two cycles of induction will be assessed using visual categorical response. The neck node measurements will be performed clinically by the treating medical oncology physician and dictated in his/her assessment note.
  * Partial response - 99%-50% decrease
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 30 | 33 | 11
Participants | 11 | 14 | 7

6. Secondary Outcome: Arms 1, 2, and 3: Anatomic Tumor Response as Assessed by CT Using RECIST 1.1 Criteria
Description: -Computed tomography (CT) scan (intravenous contrast preferred) to document and measure the extent of the primary tumor size and involved regional neck nodes. RECIST 1.1 will be used to determine response at the primary tumor site, at the involved regional neck nodes and the radiographic overall tumor response.
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 39 | 15
Participants
  Complete response | 2 | 1 | 1
  Partial response | 22 | 20 | 13

7. Secondary Outcome: Arms 1, 2, and 3: Document and Quantify Ki-67 Expression by IHC in Primary Tumor Tissue and Correlate With Clinical Primary Tumor Site Response
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Population: The data was not collected for this outcome measure.
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Arms 1, 2, and 3: Number of Participants Who Experienced a Grade 3-4 Adverse Event as Measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Compare to those observed with APF with the objective that Arm 1 will be at least 25% lower than the risk of Grade 3-4 AE's during APF (40% decreased to 30%) and Arm 2 will be at least 50% lower than the risk of Grade 3-4 AE's during APF (40% decreased to 20%).
Time Frame: 30 days after completion of treatment (estimated to be 15-25 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Nab-Paclitaxel and Cisplatin (AP) Induction: * Six weeks of nab-paclitaxel (100 mg/m2/week) and cisplatin (75 mg/m2 days 1 and 22) followed by primary tumor site (PTS) assessment
  * If complete response (CR)/partial response (PR), three more weeks of nab-paclitaxel and cisplatin followed by concurrent chemoradiation therapy (CRT)
  * If <PR, move directly to CRT if not surgical candidates.
- Arm 2: Nab-Paclitaxel (A) Induction: * Six weeks of nab-paclitaxel (100 mg/m2/week) followed by primary tumor site (PTS) assessment
  * If CR/PR, three more weeks of nab-paclitaxel followed by CRT
  * If <PR, move directly to CRT if not surgical candidates.
- Arm 3: Nab-Paclitaxel and Cisplatin (AP) Induction: * 6 weeks of nab-paclitaxel and cisplatin (days 1 & 22) followed by primary tumor site assessment
  * If CR/PR, cycle 3 of induction then 42Gy radiation, 1 dose of cisplatin or 6 doses cetuximab
  * If SD/PD: undergo surgery if candidate followed by CRT
- Arm 1 CRT: Cisplatin + Radiation Therapy: * CRT includes cisplatin which will begin 1 to 35 days after the completion of cycle 3. The first dose of cisplatin will be given during the initial 5 days of definitive radiation therapy, the second on approximately Day 22 of radiation, and the third on approximately Day 43 of radiation.
  * It is strongly recommended that intensity-modulated radiation therapy (IMRT) begin within 21 to 42 days (no later than 56 days) after the start of cycle 3. The total dose will be 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to areas considered to be an intermediate risk.
- Arm 1 & 2 ERT: Cetuximab + Radiation Therapy: * CRT includes cetuximab and will begin 1 to 35 days after completion of cycle -Cetuximab will be started 7 days before starting definitive radiation therapy. The initial loading dose of cetuximab will be 400 mg/m^2. Subsequently, cetuximab will be given weekly at a dose of 250 mg/m^2 for seven additional doses concurrently with radiation therapy.
  * It is strongly recommended that IMRT begin within 21 to 42 days (no later than 56 days) after the start of cycle 3. The total dose will be 7000 cGy in 35 fractions of 200 cGy each over 7 weeks. A dose of 6300 cGy in 35 fractions is optional and may be delivered to areas considered to be an intermediate risk.
- Arm 3 CR: Cisplatin + Radiation Therapy: * CRT includes Cisplatin and will begin 1-35 days after the completion of Cycle 3 of induction. Cisplatin will be given as 1 dose during the initial 5 days of definitive radiation therapy
  * Strongly recommended that radiation therapy begin within 28-49 days (and no later than 56 days) after the start of Cycle 3. Intensity modulated radiation therapy is to be used exclusively for this study.
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) Induction | Arm 2: Nab-Paclitaxel (A) Induction | Arm 3: Nab-Paclitaxel and Cisplatin (AP) Induction | Arm 1 CRT: Cisplatin + Radiation Therapy | Arm 1 & 2 ERT: Cetuximab + Radiation Therapy | Arm 3 CR: Cisplatin + Radiation Therapy
Number analyzed (Participants) | 40 | 40 | 15 | 39 | 35 | 15
Participants | 23 | 17 | 4 | 37 | 35 | 4

9. Secondary Outcome: Arms 1, 2, and 3: Mean Total Score as Measured by the FACT/GOG-NTX-4
Description: -The FACT/GOG-NTX-4 questionnaire has 4 questions about neuropathy (numbness/tingling in hands/feet and discomfort in hands/feet) with answers ranging from 0 (Not at all) to 4 (Very Much). The total score ranges from 0 to 16. A lower score indicates less neuropathy symptoms.
Time Frame: Baseline and one year after completion of treatment (approximately 74 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 39 | 15
score on a scale
  Baseline | 0.19 [0.02 to 0.36] | 0.38 [0.18 to 0.59] | 0.27 [0.04 to 0.57]
  End of treatment | 1.55 [1.09 to 2.01] | 0.91 [0.40 to 1.33] | 1.54 [0.90 to 2.18]

10. Secondary Outcome: Arms 1, 2, and 3: Mean Total Score as Measured by FACT-H&N
Description: -The FACT-H&N has 5 domains with 39 items including physical well-being (PWB), social/family well being (SWB), emotional well-being (EWB), functional well-being (FWB), and head & neck cancer (HNCS) with answers ranging from 0 (Not at all) to 4 (Very Much). The PWB subscale score ranges from 0-28. The SWB subscale score ranges from 0-28. The EWB subscale score ranges from 0-24. The FWB subscale score ranges from 0-28. The HNCS subscale score ranges from 0-40. To obtain the total score all subscales are added together. The total score ranges from 0-148 with a higher score indicating a better quality of life.
Time Frame: Baseline and one year after completion of treatment (approximately 74 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 39 | 15
score on a scale
  Baseline | 2.02 [1.93 to 2.11] | 1.86 [1.74 to 1.97] | 2.07 [1.94 to 2.20]
  End of treatment | 1.98 [1.89 to 2.06] | 1.82 [1.71 to 1.93] | 2.00 [1.86 to 2.15]

11. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Overall Survival (OS)
Description: OS: duration of time from date of diagnosis to late date alive or time of death from any cause.
Time Frame: Through one year after completion of treatment (approximately 74 weeks)
Population: 2 participants were excluded in Arm 3 because they received full dose radiation therapy instead of reduced dose radiation therapy.
Measure: Number; unit: percentage of particpants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of particpants | 100 | 87.50 | 92.31

12. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Overall Survival (OS)
Description: OS: duration of time from date of diagnosis to last date alive or time of death from any cause.
Time Frame: Through 2 years after completion of treatment (estimated to be 2 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 97.44 | 69.63 | 84.62

13. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Disease-free Survival (DFS)
Description: DFS: duration of time from last date of treatment to time of disease progression or death from any cause.
Time Frame: Through one year after completion of treatment (approximately 74 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 87.50 | 62.50 | 76.92

14. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Disease-free Survival (DFS)
Description: DFS: duration of time from last date of treatment to time of disease progression or death from any cause.
Time Frame: Through 2 years after completion of treatment (estimated to be 2 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 87.50 | 51.81 | 69.23

15. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Progression-free Survival (PFS)
Description: ◦PFS: duration of time from date of diagnosis to time of disease progression or death from any cause, whichever occurs first.
Time Frame: Through one year after completion of treatment (approximately 74 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 92.50 | 67.50 | 76.92

16. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Progression-free Survival (PFS)
Description: as for outcome 15
Time Frame: Through 2 years after completion of treatment (estimated to be 2 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 87.43 | 54.89 | 69.23

17. Secondary Outcome: Arm 3: Clinical Complete Response Rate as Measured by Clinical Exam at the Primary Tumor Site
Description: as for outcome 1
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Population: Only participants enrolled in Arm 3 are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 0 | 0 | 15
Participants |  |  | 9

18. Secondary Outcome: Arm 1 and Arm 3: Comparison of Response Rate
Description: -Stratified for HPV status
Time Frame: Completion of 2 cycles (approximately 6 weeks)
Population: Data was not collected for this outcome measure.
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Arm 1 and Arm 3: Comparison of the Rate of Grade 3/4 Adverse Events
Time Frame: 30 days after completion of treatment (estimated to be 15-25 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) Induction | Arm 3: Nab-Paclitaxel and Cisplatin (AP) Induction | Arm 1 CRT: Cisplatin + Radiation Therapy | Arm 3 CR: Cisplatin + Radiation Therapy
Number analyzed (Participants) | 40 | 15 | 39 | 15
Participants | 23 | 4 | 37 | 4

20. Secondary Outcome: Comparison of Median Absolute Weight Loss in Arms 2 and 3 to Arm 1
Time Frame: From start of radiation treatment through completion of radiation treatment (estimated to be 7 weeks)
Measure: Median (Full Range); unit: kilograms
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 39 | 35 | 15
kilograms | 8.4 [3.1 to 20.8] | 5.2 [4.9 to 14.6] | 7.0 [1.7 to 12.8]

21. Secondary Outcome: Comparison of Median Percent Weight Loss in Arms 2 and 3 to Arm 1
Time Frame: From start of radiation treatment through completion of radiation treatment (estimated to be 7 weeks)
Measure: Median (Inter-Quartile Range); unit: median percent of weight loss
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 15
median percent of weight loss | 9.1 [6.7 to 11.2] | 6.6 [2.6 to 8.1] | 6.7 [2.2 to 9.9]

22. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Overall Survival (OS)
Description: OS: duration of time from start of treatment to time of death from any cause
Time Frame: Up to 5 years after completion of treatment (estimated to be 5 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 77.1 | 40.5 | 68.4

23. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Progression-free Survival (PFS)
Description: ◦PFS: duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: Up to 5 years after completion of treatment (estimated to be 5 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 77.2 | 33.8 | 69.2

24. Secondary Outcome: Arms 1, 2, and 3: Kaplan-Meier Estimate of Disease-free Survival (DFS)
Time Frame: Through 5 years after completion of treatment (estimated to be 5 years and 22 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 2: Nab-Paclitaxel (A) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 40 | 13
percentage of participants | 77.2 | 32.0 | 69.2

25. Secondary Outcome: Arm 1 and Arm 3: Kaplan-Meier Estimate of Overall Survival
Time Frame: Through 5 years after completion of treatment (estimated to be 5 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 13
percentage of participants | 77.1 | 68.4

26. Secondary Outcome: Arm 1 and Arm 3: Kaplan-Meier Estimate of Disease-free Survival
Time Frame: Through 5 years after completion of treatment (estimated to be 5 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 13
percentage of participants | 77.2 | 69.2

27. Secondary Outcome: Arm 1 and Arm 3: Kaplan-Meier Estimate of Progression-free Survival
Time Frame: Through 5 years after completion of treatment (estimated to be 5 years and 22 weeks)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) + CRT | Arm 3: Nab-Paclitaxel and Cisplatin (AP) + Modified CRT
Number analyzed (Participants) | 40 | 13
percentage of participants | 77.2 | 69.2

ADVERSE EVENTS:
Time Frame: -Adverse events were collected from start of treatment through 30 days following last day of study treatment. -All-cause mortality was collected from start of treatment until completion of follow-up (up to 72 months following completion of treatment).
Description: -Participants at risk is zero for Other (Not Including Serious) Adverse Events for Arm 1 Follow-up, Arm 2 Follow-up, and Arm 3 Follow-up because adverse events were not collected in the follow-up period.
Groups:
- Arm 1: Nab-Paclitaxel+Cisplatin+CRT Follow-up; Arm 2: Nab-Paclitaxel + ERT Follow-up; Arm 3: Nab-Paclitaxel+Cisplatin+Modified CRT Follow-up: -Follow-up time period of up to 72 months post-completion of therapy
Arm/Group | Arm 1: Nab-Paclitaxel and Cisplatin (AP) Induction | Arm 2: Nab-Paclitaxel (A) Induction | Arm 3: Nab-Paclitaxel and Cisplatin (AP) Induction | Arm 1 CRT: Cisplatin + Radiation Therapy | Arm 1 & 2 ERT: Cetuximab + Radiation Therapy | Arm 3 CR: Cisplatin + Radiation Therapy | Arm 1: Nab-Paclitaxel+Cisplatin+CRT Follow-up | Arm 2: Nab-Paclitaxel + ERT Follow-up | Arm 3: Nab-Paclitaxel+Cisplatin+Modified CRT Follow-up
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/15 | 0/34 | 0/42 | 0/15 | 9/40 | 21/40 | 4/15
Serious Adverse Events (participants affected / at risk) | 6/40 | 6/40 | 2/15 | 9/34 | 6/42 | 2/15 | 0/40 | 1/40 | 1/15
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40 | 15/15 | 34/34 | 42/42 | 15/15 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Nab-Paclitaxel and Cisplatin (AP) Induction (N=40) | Arm 2: Nab-Paclitaxel (A) Induction (N=40) | Arm 3: Nab-Paclitaxel and Cisplatin (AP) Induction (N=15) | Arm 1 CRT: Cisplatin + Radiation Therapy (N=34) | Arm 1 & 2 ERT: Cetuximab + Radiation Therapy (N=42) | Arm 3 CR: Cisplatin + Radiation Therapy (N=15) | Arm 1: Nab-Paclitaxel+Cisplatin+CRT Follow-up (N=40) | Arm 2: Nab-Paclitaxel + ERT Follow-up (N=40) | Arm 3: Nab-Paclitaxel+Cisplatin+Modified CRT Follow-up (N=15)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | NA | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0 | NA | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | NA | 0 | 0
Thrombosis/embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | NA | 0 | 0
Creatinine (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | NA | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | NA | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | NA | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 1 | NA | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | NA | 0 | 0
Febrile neutropenia (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | NA | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Blood infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1 | 0
Cardiac/heart pain (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Confusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | NA | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | NA | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Throat/pharynx/larynx pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Allergic reaction - cetuximab (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Chest/thorax pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0 | 0
Death due to disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Nab-Paclitaxel and Cisplatin (AP) Induction (N=40) | Arm 2: Nab-Paclitaxel (A) Induction (N=40) | Arm 3: Nab-Paclitaxel and Cisplatin (AP) Induction (N=15) | Arm 1 CRT: Cisplatin + Radiation Therapy (N=34) | Arm 1 & 2 ERT: Cetuximab + Radiation Therapy (N=42) | Arm 3 CR: Cisplatin + Radiation Therapy (N=15) | Arm 1: Nab-Paclitaxel+Cisplatin+CRT Follow-up (N=0) | Arm 2: Nab-Paclitaxel + ERT Follow-up (N=0) | Arm 3: Nab-Paclitaxel+Cisplatin+Modified CRT Follow-up (N=0)
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 1 | 0 | 4 | 1 | NA | NA | NA
Cardiac ischemia/infarction (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Carotid artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Congestive heart failure (Cardiac disorders) | 0 | 2 | 0 | 0 | 2 | 0 | NA | NA | NA
Coronary artery disease (Cardiac disorders) | 3 | 6 | 0 | 1 | 6 | 0 | NA | NA | NA
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 11 | 5 | 0 | 8 | 11 | 1 | NA | NA | NA
Systolic murmur (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Ear pain (Ear and labyrinth disorders) | 8 | 3 | 0 | 1 | 0 | 0 | NA | NA | NA
Hearing (with baseline audiogram) (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Hearing (without monitoring program) (Ear and labyrinth disorders) | 0 | 14 | 1 | 4 | 13 | 4 | NA | NA | NA
Middle ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 3 | 1 | 0 | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 11 | 2 | 6 | 14 | 2 | 6 | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA
Corneal abrasion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Eyelid dysfunction (Eye disorders) | 2 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA
Eyelid swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA
Subconjuctival sclera hemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Vision photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Watery eyes (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 3 | 0 | NA | NA | NA
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Colon polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 14 | 14 | 8 | 12 | 16 | 4 | NA | NA | NA
Dental/teeth/periodontal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 12 | 7 | 8 | 7 | 9 | 2 | NA | NA | NA
Distension/bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 4 | 20 | 22 | 15 | NA | NA | NA
Dysgeusia (Gastrointestinal disorders) | 7 | 4 | 9 | 17 | 17 | 13 | NA | NA | NA
Dyspepsia/heartburn (Gastrointestinal disorders) | 3 | 2 | 3 | 3 | 1 | 0 | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 20 | 25 | 6 | 20 | 29 | 13 | NA | NA | NA
GERD (Gastrointestinal disorders) | 6 | 4 | 0 | 7 | 6 | 0 | NA | NA | NA
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Mucositis oral (Gastrointestinal disorders) | 4 | 0 | 1 | 26 | 34 | 15 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 18 | 14 | 12 | 24 | 16 | 9 | NA | NA | NA
Odynophagia (Gastrointestinal disorders) | 4 | 3 | 0 | 4 | 6 | 0 | NA | NA | NA
Oral cavity hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Oral cavity pain (Gastrointestinal disorders) | 2 | 2 | 0 | 8 | 4 | 1 | NA | NA | NA
Oropharyngeal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Salivary gland changes/saliva (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | NA | NA | NA
Stoma hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA
Stomach stricture (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA
Stomatitis (oral cavity) (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Teeth (dental caries) (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 2 | 5 | 1 | 13 | 7 | 6 | NA | NA | NA
Cervical adenopathy (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Face pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Fatigue (General disorders) | 24 | 21 | 10 | 29 | 26 | 13 | NA | NA | NA
Fever (General disorders) | 4 | 2 | 2 | 6 | 4 | 0 | NA | NA | NA
Flu-like syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA
General edema (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA
Head and neck edema (General disorders) | 3 | 3 | 1 | 0 | 4 | 1 | NA | NA | NA
Limb edema (General disorders) | 5 | 8 | 1 | 6 | 12 | 2 | NA | NA | NA
Obesity (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Pain - NOS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Pain in bottoms of feet (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Rigors/chills (General disorders) | 1 | 3 | 0 | 4 | 3 | 0 | NA | NA | NA
Agammaglobulinemia (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Allergic reaction - cetuximab (Immune system disorders) | 0 | 0 | 0 | 0 | 5 | 0 | NA | NA | NA
Bacteremia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Blood infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA
Catheter related infection (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 0 | NA | NA | NA
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Febrile neutropenia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | NA | NA | NA
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Oral thrush (Infections and infestations) | 0 | 1 | 0 | 4 | 3 | 2 | NA | NA | NA
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | NA | NA | NA
Shingles (Infections and infestations) | 1 | 0 | 0 | 0 | 7 | 0 | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 4 | 0 | 0 | 0 | 0 | NA | NA | NA
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Upper airway NOS infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 1 | 4 | 0 | NA | NA | NA
Viral hepatitis (Infections and infestations) | 0 | 5 | 0 | 0 | 2 | 0 | NA | NA | NA
Viral respiratory infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Bruising (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA
Dermatitis - chemoradiation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 21 | 33 | 12 | NA | NA | NA
Dermatitis - chemotherapy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 5 | 0 | NA | NA | NA
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
G-tube pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Induration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0 | NA | NA | NA
ALT (Investigations) | 7 | 8 | 1 | 6 | 8 | 0 | NA | NA | NA
AST (Investigations) | 4 | 9 | 1 | 3 | 8 | 1 | NA | NA | NA
Alkaline phosphatase (Investigations) | 4 | 6 | 1 | 5 | 7 | 1 | NA | NA | NA
Cardiac troponin I (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Creatinine (Investigations) | 9 | 14 | 2 | 20 | 11 | 4 | NA | NA | NA
Hemoglobin (Investigations) | 40 | 35 | 15 | 34 | 35 | 15 | NA | NA | NA
Hyperbilirubinemia (Investigations) | 0 | 1 | 1 | 0 | 2 | 0 | NA | NA | NA
Hypercholesterolemia (Investigations) | 3 | 2 | 0 | 2 | 3 | 0 | NA | NA | NA
INR (Investigations) | 2 | 5 | 1 | 7 | 11 | 2 | NA | NA | NA
Leukocytes (Investigations) | 27 | 25 | 12 | 30 | 11 | 8 | NA | NA | NA
Lymphopenia (Investigations) | 24 | 25 | 8 | 34 | 35 | 12 | NA | NA | NA
Neutropenia (ANC) (Investigations) | 27 | 21 | 13 | 26 | 5 | 4 | NA | NA | NA
PTT (Investigations) | 2 | 2 | 0 | 2 | 6 | 0 | NA | NA | NA
Platelets (Investigations) | 16 | 3 | 1 | 23 | 7 | 6 | NA | NA | NA
Weight loss (Investigations) | 8 | 9 | 4 | 29 | 27 | 8 | NA | NA | NA
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Anorexia (Metabolism and nutrition disorders) | 8 | 7 | 3 | 8 | 17 | 4 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2 | 12 | 6 | 6 | NA | NA | NA
Diabetes (Metabolism and nutrition disorders) | 5 | 9 | 2 | 4 | 11 | 2 | NA | NA | NA
GFR (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | NA | NA | NA
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 2 | 3 | 0 | NA | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 9 | 1 | 9 | 9 | 1 | NA | NA | NA
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 10 | 2 | 7 | 5 | 1 | NA | NA | NA
Hyperlipidemia (Metabolism and nutrition disorders) | 3 | 3 | 4 | 3 | 3 | 4 | NA | NA | NA
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 5 | 0 | NA | NA | NA
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 3 | 0 | NA | NA | NA
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 12 | 1 | 20 | 26 | 2 | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 6 | 0 | 16 | 17 | 2 | NA | NA | NA
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 1 | 0 | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 5 | 5 | 2 | 16 | 14 | 1 | NA | NA | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 6 | 2 | 9 | 11 | 3 | NA | NA | NA
Hyponatremia (Metabolism and nutrition disorders) | 11 | 14 | 2 | 24 | 16 | 6 | NA | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 7 | 7 | 1 | NA | NA | NA
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Armpit pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 2 | 2 | 0 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 3 | 2 | 1 | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Extremity muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Extremity/limb pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 4 | 3 | 1 | NA | NA | NA
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA
Joint pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 3 | 1 | 1 | NA | NA | NA
Joint-function (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA
Lower extremity muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Lower limb generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 0 | 3 | 6 | 0 | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Soft tissue necrosis - neck (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Trismus (Musculoskeletal and connective tissue disorders) | 7 | 6 | 0 | 6 | 6 | 2 | NA | NA | NA
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 8 | 6 | 3 | 5 | 2 | NA | NA | NA
Anoxic brain injury (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Apnea (Nervous system disorders) | 4 | 1 | 2 | 3 | 1 | 2 | NA | NA | NA
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
CNS ischemia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA
Confusion (Nervous system disorders) | 1 | 0 | 1 | 2 | 2 | 0 | NA | NA | NA
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Dizziness (Nervous system disorders) | 7 | 4 | 3 | 6 | 7 | 6 | NA | NA | NA
Dysphasia (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 4 | 3 | 3 | 2 | 4 | 1 | NA | NA | NA
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Parkinson's disease (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | NA | NA | NA
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA
Anxiety (Psychiatric disorders) | 7 | 9 | 3 | 9 | 7 | 6 | NA | NA | NA
Depression (Psychiatric disorders) | 1 | 5 | 1 | 6 | 5 | 2 | NA | NA | NA
Insomnia (Psychiatric disorders) | 5 | 4 | 1 | 1 | 3 | 2 | NA | NA | NA
OCD (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Psychosis (bipolar disorder) (Psychiatric disorders) | 0 | 2 | 0 | 0 | 2 | 0 | NA | NA | NA
Sensory neuropathy (Psychiatric disorders) | 6 | 11 | 4 | 14 | 6 | 9 | NA | NA | NA
BPH (Renal and urinary disorders) | 1 | 2 | 0 | 1 | 1 | 0 | NA | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Chronic renal insufficiency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | NA | NA | NA
Kidney stone (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 0 | 0 | NA | NA | NA
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Polycistic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Proteinuria (Renal and urinary disorders) | 2 | 4 | 0 | 7 | 7 | 0 | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 1 | 0 | NA | NA | NA
Urinary frequency (Renal and urinary disorders) | 1 | 3 | 0 | 1 | 1 | 0 | NA | NA | NA
Urinary hemorrhage (Renal and urinary disorders) | 2 | 3 | 0 | 2 | 6 | 0 | NA | NA | NA
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0 | 7 | 2 | 0 | NA | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | NA | NA | NA
Bronchospasm/wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 3 | 0 | NA | NA | NA
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 0 | 0 | 8 | 0 | NA | NA | NA
Chest/thorax NOS pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Chronic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 1 | 16 | 10 | 1 | NA | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 1 | 4 | 6 | 1 | NA | NA | NA
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1 | 0 | 0 | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Larynx hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Nose hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 1 | 1 | NA | NA | NA
Nose pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Pharynx hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
RSV (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Respiratory tract NOS hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | NA | NA | NA
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA
Throat/pharynx/larynx pain (Respiratory, thoracic and mediastinal disorders) | 13 | 12 | 1 | 17 | 14 | 1 | NA | NA | NA
Trachea hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 16 | 22 | 1 | 14 | 23 | 2 | NA | NA | NA
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 14 | 4 | 20 | 21 | 4 | NA | NA | NA
Boil (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Cystic lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4 | 5 | 2 | NA | NA | NA
Ecchymoses (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 7 | 3 | 0 | NA | NA | NA
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 2 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | NA | NA | NA
Rash unexplained (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 | 10 | 3 | 5 | 5 | 0 | NA | NA | NA
Rash: acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 18 | 0 | NA | NA | NA
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Sweating (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 1 | 3 | 0 | NA | NA | NA
Ungual infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA
Hypertension (Vascular disorders) | 30 | 30 | 7 | 25 | 26 | 6 | NA | NA | NA
Hypotension (Vascular disorders) | 3 | 0 | 1 | 2 | 1 | 1 | NA | NA | NA
Peripheral vascular disease (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA
Thrombosis/embolism (Vascular disorders) | 4 | 1 | 0 | 4 | 4 | 1 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT02573493/Prot_SAP_000.pdf